CLINICAL TRIAL: NCT03880760
Title: The Effect of Probiotics on Type 1 Diabetes Mellitus in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chung-Hsing Wang, Attending physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH107-REC2-036
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1DM; Autoimmune diseases; Microbiota; Probiotics
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Probiotics or placebo group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics capsule (Experimental): Taking 1 L. johnsonii MH-68, B. animalis subsp. lactis CP-9 and L. salivarius AP-32 mix probiotics capsule twice a day before meals for six months.
  Interventions: Other: L. johnsonii MH-68, B. animalis subsp. lactis CP-9 and L. salivarius AP-32
- Placebo capsule (Placebo Comparator): Taking 1 placebo capsule twice a day before meals for six months.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: L. johnsonii MH-68, B. animalis subsp. lactis CP-9 and L. salivarius AP-32 — Taking 1 L. johnsonii MH-68, B. animalis subsp. lactis CP-9 and L. salivarius AP-32 mix probiotics capsule twice a day before meals for six months.
  Arms: Probiotics capsule
Other: Placebo — Taking 1 placebo capsule twice a day before meals for six months.
  Arms: Placebo capsule

SUMMARY:
In this study, investigators try to administer probiotics (Lactobacillus salivarius + Lactobacillus johnsonii + Bifidobacterium lactis from glac biotech Co., Ltd.) to children T1DM patients for 6 months to observe if the inhibition effect of T1DM animal model could be discerned in a short-term period from both change of serum cytokines and beta cells insulin secretion ability.

DETAILED DESCRIPTION:
Type 1 (insulin-dependent) Diabetes Mellitus (T1DM) is among the most well studied organ-specific autoimmune diseases which approximately 75% of newly diagnosed DM patients acquire this type before the age of 18. T1DM is well known for as the consequence of selective destruction of pancreatic insulin-producing beta cells within the islets of Langerhans. Basically, autoimmune reactions against beta cells may come from activation of the immune system in genetically susceptible individuals triggered by environmental factors that bear epitopes similar to those expressed by the beta cells. Several mechanisms such as molecular mimicry, metabolic stress on beta cells, cryptic epitope exposure and costimulatory molecule upregulation have been proposed but none of them could be solely responsible for the pathogenesis of T1DM. Recently, T1DM has been considered a consequence of dysregulated or over-activation of immune responses in genetically predisposed individuals, similar to other autoimmune diseases.

The rapid increase in the incidence of T1DM in developed countries including Taiwan during recent decades refers to the role of environmental factors in this disease. Candidate environmental factors influencing T1DM include various microbial and food components encountered at mucosal surfaces as well as gut mucosal parameters such as gut permeability. However, difficulty exists in characterizing the environmental factors and mechanisms in T1DM because of their complexity of interaction, the long lag period between the induction of disease trigger factors and the clinical onset of the disease. Environmental factors in T1DM seem to prevent full penetration of the disease rather than trigger it. It had been reported that high diabetes incidence in germ-free mice and an involvement of innate immune mechanisms in the disease. In this study, investigators try to administer probiotics (Lactobacillus salivarius + Lactobacillus johnsonii + Bifidobacterium lactis from glac biotech Co., Ltd.) to children T1DM patients for 6 months to see if the inhibition effect of T1DM animal model could be discerned in a short-term period from both change of serum cytokines and beta cells insulin secretion ability.

Subjects will collect blood before the test and every 3 months after the test for total 4 times. Each time the collected blood volume is about 5~8cc. A part of the blood sample will be given to the Department of laboratory medicine for the detection of hemoglobin A1c (HbA1c) and fasting blood glucose, and the other part will be centrifuged to separate serum. The serum macrophage inflammatory proteins-1beta (MIP-1β), regulated on activation, normal T cell expressed and secreted (RANTES), interleukin-8 (IL-8), interleukin-17 (IL-17), tumor necrosis factor alpha (TNF-α) and transforming growth factor beta1 (TGF-β1) concentrations will be measured by ELISA.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 to 18 years old.
2. T1DM patients confirmed by glucagon tests and/or presence of autoantibody(ies).

Exclusion Criteria:

1. Significant cardiac, renal and hepatic disease.
2. The physician diagnosed the immunodeficiency or the immune function was low.
3. Currently using probiotics supplements or had ever taken probiotics for more than one month.
4. Currently using antibiotics or gastrointestinal medicine.
5. Ever allergic reaction(s) to probiotics or prebiotics regimen.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change in percentage of HbA1c | From date of first blood draw after entering the trial until the date of third blood draw, assessed up to 6 months.
  Subjects will draw blood once before the test. During the test, every 3 months will draw blood to 6th month, each time the blood volume is about 5 ~ 8cc to detect HbA1c and other blood biochemical values.
Change in concentration of blood glucose (AC) | From date of first blood draw after entering the trial until the date of third blood draw, assessed up to 6 months.
  The study will require subject to record their own daily fasting blood glucose.

SECONDARY OUTCOMES:
Change in concentration of MIP-1β | From date of first blood draw after entering the trial until the date of third blood draw, assessed up to 6 months.
  Serum was isolated by extra blood draw, serum MIP-1β (pg/ml) concentrations were measured from first blood draw to third blood draw by ELISA.
Change in concentration of RANTES | From date of first blood draw after entering the trial until the date of third blood draw, assessed up to 6 months.
  Serum was isolated by extra blood draw, serum RANTES (pg/ml) concentrations were measured from first blood draw to third blood draw by ELISA.
Change in concentration of IL-8 | From date of first blood draw after entering the trial until the date of third blood draw, assessed up to 6 months.
  Serum was isolated by extra blood draw, serum IL-8 (pg/ml) concentrations were measured from first blood draw to third blood draw by ELISA.
Change in concentration of IL-17 | From date of first blood draw after entering the trial until the date of third blood draw, assessed up to 6 months.
  Serum was isolated by extra blood draw, serum IL-17 (pg/ml) concentrations were measured from first blood draw to third blood draw by ELISA.
Change in concentration of TNF-α | From date of first blood draw after entering the trial until the date of third blood draw, assessed up to 6 months.
  Serum was isolated by extra blood draw, serum TNF-α (pg/ml) concentrations were measured from first blood draw to third blood draw by ELISA.
Change in concentration of TGF-β1 | From date of first blood draw after entering the trial until the date of third blood draw, assessed up to 6 months.
  Serum was isolated by extra blood draw, serum TGF-β1 (pg/ml) concentrations were measured from first blood draw to third blood draw by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-chih Lin, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Wang CH, Yen HR, Lu WL, Ho HH, Lin WY, Kuo YW, Huang YY, Tsai SY, Lin HC. Adjuvant Probiotics of Lactobacillus salivarius subsp. salicinius AP-32, L. johnsonii MH-68, and Bifidobacterium animalis subsp. lactis CP-9 Attenuate Glycemic Levels and Inflammatory Cytokines in Patients With Type 1 Diabetes Mellitus. Front Endocrinol (Lausanne). 2022 Mar 1;13:754401. doi: 10.3389/fendo.2022.754401. eCollection 2022. PMID 35299968